CLINICAL TRIAL: NCT07406139
Title: A Multicenter, Prospective, Single-arm Exploratory Study of Prothrombin Complex Concentrate in the Treatment of Bleeding Episodes in Patients With Hemophilia A With Inhibitors
Brief Title: PCC Treatment for Hemophilia Patients With Inhibitor（2022PCC-A）
Acronym: 2022PCC-A
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: North China University of Science and Technology (Other); The Second Affiliated Hospital of Kunming Medical University (Other); The Second People's Hospital of Anhui Province (Other); Children's Hospital of Chongqing Medical University (Other); Union Hospital, Affiliated to Fujian Medical University (Unknown); The First Affiliated Hospital of Xiamen University (Other); First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022048
Record Dates: First submitted 2025-11-20; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Hemophilia; Inhibitors
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PCC treatment (Experimental)
  Interventions: Drug: PCC

INTERVENTIONS:
Drug: PCC — On-demand PCC therapy during bleeding episodes. The recommended dose was 50 IU/kg per infusion, administered every 8-12 hours, with a maximum total daily dose not exceeding 150 IU/kg.

SUMMARY:
This study is a multicenter, prospective, single-arm exploratory clinical trial designed to evaluate the efficacy and safety of prothrombin complex concentrate (PCC) in the treatment of bleeding episodes in patients with hemophilia A with inhibitors. All participants received on-demand PCC therapy during bleeding episodes, with dosing adjusted by investigators according to the type of bleeding. The recommended dose was 50 IU/kg per infusion, administered every 8-12 hours, with a maximum total daily dose not exceeding 150 IU/kg. If no effective hemostasis was achieved within 24 hours, investigators could decide to add other hemostatic agents or switch to alternative treatments.

DETAILED DESCRIPTION:
Hemophilia A is a severe and common hereditary bleeding disorder caused by a deficiency of coagulation factor VIII (FVIII). Recurrent bleeding episodes, if not treated promptly, can lead to joint deformities or pseudotumor formation and may even be life-threatening in severe cases. In recent years, with the widespread use of plasma-derived and recombinant FVIII products, the management of hemophilia A has made significant progress. Increasing numbers of patients are now receiving prophylactic care and appropriate surgical interventions, resulting in substantial improvements in quality of life.

However, the incidence of inhibitors in hemophilia A has been rising. Approximately 30% of patients with severe hemophilia A and 3-13% of those with non-severe disease develop inhibitors. The presence of inhibitors neutralizes FVIII activity, rendering FVIII replacement therapy ineffective, thereby increasing the risk of life-threatening bleeding and contributing to severe joint damage. Activated prothrombin complex concentrate (aPCC) and recombinant activated factor VII (rFVIIa) are two commonly used "bypassing agents" worldwide. These agents achieve hemostasis by generating thrombin through pathways that bypass the need for FVIII or FIX activation.

According to Cochrane systematic reviews, both aPCC and rFVIIa achieve hemostatic efficacy rates above 80%, demonstrate similar tolerability, and have a low incidence of thrombotic complications. However, since aPCC is not available in China and rFVIIa is costly, prothrombin complex concentrate (PCC) is generally used as an alternative. The 2020 Chinese Guidelines for the Management of Hemophilia recommend PCC and rFVIIa as bypassing options for patients with high-titer inhibitors (>5 BU/mL), those who fail immune tolerance induction (ITI), or those who experience bleeding during ITI therapy.

PCC is a plasma-derived concentrate obtained from pooled plasma of healthy donors, containing mainly vitamin K-dependent coagulation factors II, VII, IX, and X. It is categorized as either a four-factor PCC (containing therapeutic levels of FVII, as well as anticoagulant proteins C and S) or a three-factor PCC (with lower levels of FVII and anticoagulant proteins). Four-factor PCC can enhance thrombin generation directly or indirectly on platelet surfaces, with elevated FVII levels likely being a key contributor to its procoagulant effect. Meanwhile, the presence of balancing anticoagulant proteins C and S may help mitigate excessive coagulation and reduce thrombotic risk.

To date, no prospective clinical study has been conducted in China to evaluate the efficacy and safety of PCC in the management or prophylaxis of bleeding in hemophilia A patients with inhibitors; available data are limited to retrospective analyses and case reports. Considering the current situation in China, a prospective evaluation of the efficacy and safety of four-factor PCC for hemostasis in hemophilia A patients with inhibitors is of great importance, as it can provide more objective and scientific evidence for clinical decision-making. In addition, since patient-specific factors, the mechanisms of bypassing agents, and pharmacokinetic variability can all lead to differing treatment responses, this study also incorporates thrombin generation assay (TGA) testing to assess individual patient responses and provide further objective data supporting the hemostatic efficacy of four-factor PCC.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with hemophilia A with inhibitors. For high-responding patients (those who have previously had an inhibitor titer >5 BU), the inhibitor titer at enrollment must be >0.6 BU;
2. Age between 12 and 65 years;
3. At least three joint bleeding episodes within the past six months;
4. Signed informed consent form.

Exclusion Criteria:

1. Presence of other congenital or acquired bleeding disorders;
2. Liver function tests (ALT, AST) >2.5 times the upper limit of normal, or renal function tests (BUN, Cr) >1.5 times the upper limit of normal;
3. Currently receiving immune tolerance induction (ITI) therapy with an inhibitor titer <5 BU;
4. History of thrombotic events;
5. Known history of drug allergy, asthma, urticaria, or other allergic conditions;
6. Deemed unsuitable for study participation by the investigator.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Efficacy of prothrombin complex concentrate (PCC) in the treatment of bleeding episodes in patients with hemophilia A with inhibitors. | From enrollment to the end of treatment at 24 hours
  Hemostatic Efficacy Rate:
  Bleeding symptoms were evaluated at 8 hours and 24 hours after treatment. The assessment of hemostatic response included four categories: excellent, good, moderate, and ineffective.

SECONDARY OUTCOMES:
To evaluate the improvement score of bleeding symptoms and signs within 24 hours after the first infusion of prothrombin complex concentrate (PCC) for each bleeding episode in patients with hemophilia A with inhibitors. | From enrollment to the end of treatment at 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of haematology and Blood diseases hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months 36 months after study completion.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months to 36 months after study completion
Access Criteria: Upon request to PI